CLINICAL TRIAL: NCT06447610
Title: Lateral Arm Free Flap: a Useful Flap in the Maxillo-facial Surgeon's Therapeutic Armory, Case Series
Status: Completed | Type: Observational
Sponsor: CHUV chirurgie orale et maxillofaciale (Other)
Responsible Party: Sponsor
Other Study IDs: lateral arm 1
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Reconstructive Surgery
Keywords: Free flaps; Reconstructive surgery; Microvascular surgery; maxillofacial surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lateral arm free flap — In this study, we present a case series of 8 patients operated for a maxillo-facial defect with a lateral arm free flap.

SUMMARY:
Lateral arm free flap harvesting has been well described, it however remains underused compared to other free flaps such as radial forearm and anterolateral thigh free flap. Due to its easy harvesting, low donor site morbidity, versatility as well as useful possibilities of modifications it should be considered more often as valuable reconstruction option in head and neck defect. With this publication we want to describe the operative technique, illustrate it with postoperative pictures and describe the outcome with 8 of our cases operated at University Hospital In Lausanne, Switzerland.

The aim of this study is to be a useful tool for young surgeons and demonstrate the advantages of this useful flap in head and neck reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* operated between 01 january 2021 and 12 december 2022
* lateral arm free flap operation for primary or secondary cervicofacial reconstruction
* written informed consent

Exclusion Criteria:

* minor patients
* no written informed consent

Ages: 52 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 2021 and 2022, 8 patients (1 woman and 7 men) underwent reconstruction with a lateral arm free flap in Lausanne, Switzerland (Table 1). Their ages ranged from 52 to 87 years, with a mean age of 65.25 years. The reconstruction site varied from the exenterated orbita for two patients, internal cheek for two patients, retromolar mandible, palate, mouth floor and frontotemporal each for one patient. Reconstruction was done in all patients for oncologic reason. Six patients received primary reconstruction during the same surgery as the tumorectomy and for two patients' reconstruction was done in a second surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Flap complication | 01.01.2021-12.01.2022
  Description of free flap outcome: revision, complete or partial survival

SECONDARY OUTCOMES:
Patient complication | 01.01.2021-12.01.2022
  general complcation such as cardiac, pulmonary, neurologic complcation
oral food intke | 01.01.2021-12.01.2022
  days after surgery when oral food intake is allowed
revision of anastomoses | 01.01.2021-12.01.2022
  secondary look for patency of anastomoses because of free flap suffering

CONTACTS AND LOCATIONS:
Overall Officials: Laurence May, MD, Principal Investigator — CHUV; oral and maxillofacial surgery , Lausanne, Switzerland
Locations (1):
- CHUV oral and maxillofacial surgery, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No